CLINICAL TRIAL: NCT03516279
Title: Phase II Study of Adding the Anti-PD-1 Pembrolizumab to Tyrosine Kinase Inhibitors in Patients With Chronic Myeloid Leukemia and Persistently Detectable Minimal Residual Disease
Brief Title: Pembrolizumab and Dasatinib, Imatinib Mesylate, or Nilotinib in Treating Patients With Chronic Myeloid Leukemia and Persistently Detectable Minimal Residual Disease
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EA9171; NCI-2017-02161 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA9171 (Other: ECOG-ACRIN Cancer Research Group); EA9171 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2018-04-24; First posted 2018-05-04 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Chronic Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Minimal Residual Disease
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Neoplasm, Residual | interventions — Dasatinib; Imatinib Mesylate; nilotinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (pembrolizumab, dasatinib, imatinib, nilotinib) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1 and dasatinib, imatinib mesylate, or nilotinib PO as clinically indicated per the treating physician. Treatment repeats every 21 days for up to 18 courses in the absence of disease progression or unacceptable toxicity. Patients with detectable MRD after course 18 continue pembrolizumab and dasatinib, imatinib mesylate, or nilotinib every 21 days for up to an additional 18 courses in the absence of disease progression or unacceptable toxicity. Patients with UMRD at any time before course 18 discontinue pembrolizumab after course 18 and continue dasatinib, imatinib mesylate, or nilotinib every 21 days for up to an additional 18 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Dasatinib; Drug: Imatinib Mesylate; Other: Laboratory Biomarker Analysis; Drug: Nilotinib; Biological: Pembrolizumab

INTERVENTIONS:
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Sprycel
Drug: Imatinib Mesylate — Given PO
  Other Names: CGP 57148; CGP57148B; Gleevec; Glivec; STI 571; STI-571; STI571
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Nilotinib — Given PO
  Other Names: AMN 107; Tasigna
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well pembrolizumab and dasatinib, imatinib mesylate, or nilotinib work in treating patients with chronic myeloid leukemia and persistent detection of minimal residual disease, defined as the levels of a gene product called bcr-abl in the blood. Monoclonal antibodies, such as pembrolizumab, may interfere with the ability of cancer cells to grow and spread. Dasatinib, imatinib mesylate, and nilotinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving pembrolizumab and dasatinib, imatinib mesylate, or nilotinib may work better in treating patients with chronic myeloid leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the proportion of chronic myelogenous leukemia (CML) patients on stable-dose tyrosine kinase inhibitor (TKI) who convert to undetectable minimal residual disease (UMRD) (molecular response [MR]^4.5) during or within 2 years of initiating pembrolizumab therapy.

SECONDARY OBJECTIVES:

I. Among patients who have converted to UMRD (MR^4.5), assess the proportion of CML patients who maintain UMRD for 6 months and 12 months.

II. Among patients who have converted to UMRD (MR^4.5), assess the proportion of CML patients who discontinue their TKI.

III. Among patients who have converted to UMRD (MR^4.5), assess the proportion of CML patients who are UMRD and TKI-free at 2 years from first determined UMRD.

IV. Assess the proportion of CML patients who develop grade 3 or 4 immune related adverse events related to pembrolizumab treatment during the first 2 years after registration (not including grade 3 events that respond to corticosteroids and improve to grade 1 or less within 4 weeks).

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1 and dasatinib, imatinib mesylate, or nilotinib orally (PO) as clinically indicated per the treating physician. Treatment repeats every 21 days for up to 18 courses in the absence of disease progression or unacceptable toxicity. Patients with detectable MRD after course 18 continue pembrolizumab and dasatinib, imatinib mesylate, or nilotinib every 21 days for up to an additional 18 courses in the absence of disease progression or unacceptable toxicity. Patients with UMRD at any time before course 18 discontinue pembrolizumab after course 18 and continue dasatinib, imatinib mesylate, or nilotinib every 21 days for up to an additional 18 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 6 years from the date of registration.

ELIGIBILITY:
Inclusion Criteria:

* PREREGISTRATION (STEP 0): Patient has pathologically-confirmed chronic phase-CML on a first line TKI and must meet the following criteria:

  * The patient has to be on first-line TKI therapy (the same TKI) for at least 2 years prior to pre-registration
  * Has been in MMR (i.e. MR^3) but still have detectable BCR-ABL transcript by a standard real-time quantitative polymerase chain reaction (RQ-PCR) assay with a limit of detection (sensitivity) of 4.5 for at least 12 months from the first documentation of the MMR
  * Patient has not achieved MR^4.5 (complete molecular remission [CMR]) within the time of initiation of TKI therapy and pre-registration
* PREREGISTRATION (STEP 0): Patient must be scheduled to undergo a standard of care bone marrow biopsy within 7 days of step 0 registration
* PREREGISTRATION (STEP 0): Peripheral blood must be collected for submission to Fred Hutchinson Cancer Research Center for central assessment of the establishment of BCR/ABL status to confirm patient?s eligibility for registration to Step 1; Fred Hutchinson will forward results within 1-2 business days of receipt of the peripheral blood to the submitting institution
* REGISTRATION TO TREATMENT (STEP 1): Institution has received central BCR-ABL test results confirming MRD positive status
* REGISTRATION TO TREATMENT (STEP 1): Patients have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* REGISTRATION TO TREATMENT (STEP 1): No active hemolytic anemia requiring immunosuppressive therapy or other pharmacologic treatment; patients who have a positive Coombs test but no evidence of hemolysis are NOT excluded from participation
* REGISTRATION TO TREATMENT (STEP 1): No current use of corticosteroids; EXCEPTION: Low doses of steroids (< 10 mg of prednisone or equivalent dose of other steroid) used for treatment of non-hematologic medical condition (e.g. chronic adrenal insufficiency) is permitted
* REGISTRATION TO TREATMENT (STEP 1): No other active primary malignancy (other than non-melanomatous skin cancer or carcinoma in situ of the cervix) requiring treatment or limiting expected survival to =< 2 years

  * NOTE: If there is a history of prior malignancy, they must not be receiving other specific treatment (other than hormonal therapy for their cancer)
* REGISTRATION TO TREATMENT (STEP 1): Women must not be pregnant or breastfeeding; patients must also not expect to conceive or father children from the time of registration, while on study treatment, and continue for 120 days after the last dose of study treatment; all females of childbearing potential must have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of pembrolizumab; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required; a female of childbearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* REGISTRATION TO TREATMENT (STEP 1): Women of childbearing potential and sexually active males must use an accepted and effective method of contraception or to abstain from sexual from time of registration, while on study treatment, and continue for 120 days after the last dose of study treatment
* REGISTRATION TO TREATMENT (STEP 1): Patients must have been on a stable dose of the TKI for the last 3 months prior to pre-registration
* REGISTRATION TO TREATMENT (STEP 1): Patient may not be currently participating and receiving study therapy or have participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* REGISTRATION TO TREATMENT (STEP 1): Patient must not have a diagnosis of immunodeficiency or be receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of treatment
* REGISTRATION TO TREATMENT (STEP 1): Patient must not have a known history of active TB (Bacillus Tuberculosis)
* REGISTRATION TO TREATMENT (STEP 1): Patient must not have a history of hypersensitivity to pembrolizumab or any of its excipients
* REGISTRATION TO TREATMENT (STEP 1): Patient must not have received a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study registration or have not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* REGISTRATION TO TREATMENT (STEP 1): Patient must not have had prior chemotherapy, targeted small molecule therapy (aside from imatinib, dasatinib, or nilotinib), or radiation therapy within 2 weeks prior to study registration; patients also must have recovered from all adverse events due to a previously administered agent

  * Note: Patients with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
* REGISTRATION TO TREATMENT (STEP 1): Patients who have received major surgery must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* REGISTRATION TO TREATMENT (STEP 1): Patient must not have a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* REGISTRATION TO TREATMENT (STEP 1): Patient must not have known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of protocol treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to protocol treatment; this exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
* REGISTRATION TO TREATMENT (STEP 1): Patient must not have active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* REGISTRATION TO TREATMENT (STEP 1): Patient must not have known history of, or any evidence of active, non-infectious pneumonitis
* REGISTRATION TO TREATMENT (STEP 1): Patient must not have an active infection requiring systemic therapy
* REGISTRATION TO TREATMENT (STEP 1): Patient must not have a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* REGISTRATION TO TREATMENT (STEP 1): Patient must not have known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* REGISTRATION TO TREATMENT (STEP 1): Patient must not have received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent
* REGISTRATION TO TREATMENT (STEP 1): Patients who are Human Immunodeficiency Virus (HIV) positive are eligible if they have undetectable HIV viral load and CD4+ T-cell count ≥ 250/mm3.
* REGISTRATION TO TREATMENT (STEP 1): Patients with a known positive test for Hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection might be enrolled if the viral load by PCR is undetectable with/without active treatment.
* REGISTRATION TO TREATMENT (STEP 1): Patients must not have known history of hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive).
* REGISTRATION TO TREATMENT (STEP 1): Patient must not have received a live vaccine within 30 days of planned start of study therapy

  * NOTE: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed
* REGISTRATION TO TREATMENT (STEP 1): Absolute neutrophil count (ANC) >= 1,500 /mcL, within 14 days prior to first dose of pembrolizumab
* REGISTRATION TO TREATMENT (STEP 1): Platelet count >= 100,000 /mcL, within 14 days prior to first dose of pembrolizumab
* REGISTRATION TO TREATMENT (STEP 1): Hemoglobin (Hgb) >= 9 g/dL OR >= 5.6 mmol/L without transfusion of erythropoietin (EPO) dependency, within 14 days prior to first dose of pembrolizumab
* REGISTRATION TO TREATMENT (STEP 1): Serum creatinine =< 1.5 X upper limit of normal (ULN) OR creatinine clearance (per institutional standards) >= 60 mL/min for patient with creatinine levels > 1.5 X ULN, within 14 days prior to first dose of pembrolizumab
* REGISTRATION TO TREATMENT (STEP 1): Serum total bilirubin =< 1.5 X ULN OR direct bilirubin

  =< ULN for subjects with total bilirubin levels > 1.5 X ULN, within 14 days prior to first dose of pembrolizumab
* REGISTRATION TO TREATMENT (STEP 1): Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases, within 14 days prior to first dose of pembrolizumab
* REGISTRATION TO TREATMENT (STEP 1): Patients should not be receiving concomitant strong CYP3A4 inducers or inhibitors ≤ 7 days prior to registration due to their potential to effect the activity or pharmacokinetics of study agents and/or QT interval prolongation toxicity. Should treatment with any of these agents be required, consult with study chair.
* REGISTRATION TO TREATMENT (STEP 1): Patients should not have received prior allogeneic transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-06-26 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2031-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients on tyrosine kinase inhibitor (TKI) who convert to undetectable minimal residual disease (UMRD) | Up to 2 years of initiating pembrolizumab
  Will be reported with exact confidence intervals. The binomial test will be used to test the null hypothesis that this proportion is 0.2 with the alternative hypothesis being that this proportion is greater than 0.2.

SECONDARY OUTCOMES:
Proportion of patients who maintain UMRD for 6 months | Up to 6 years
  Will be assessed among patients who achieve UMRD within two years of initiating pembrolizumab. The proportions will be reported with exact confidence intervals.
Proportion of patients who maintain UMRD for 6 and 12 months | Up to 6 years
  Will be assessed among patients who achieve UMRD within two years of initiating pembrolizumab. The proportions will be reported with exact confidence intervals.
Proportion of patients who meet the criteria for discontinuing TKI | Up to 6 years
  Will be assessed among patients who achieve and maintain UMRD within two years of initiating pembrolizumab. The proportions will be reported with exact confidence intervals.
Proportion of patients who maintain UMRD for 2 years after first achieving UMRD | Up to 6 years
  Will be assessed among patients who have converted to UMRD (molecular response [MR]^4.5) and discontinued TKI. The proportions will be reported with exact confidence intervals.
Proportion of patients who develop grade 3 or 4 immune related adverse events (not including grade 3 events that respond to corticosteroids and improve to grade 1 or less within 4 weeks) | Up to 6 years
  Will be tabulated based on grade Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Amer Zeidan, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (291):
- United States (291):
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - CARTI Cancer Center, Little Rock, Arkansas
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Mercy Cancer Center, Merced, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - BASS Medical Group - Lennon, Walnut Creek, California
  - Woodland Memorial Hospital, Woodland, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Beebe South Coastal Health Campus, Frankford, Delaware
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Saint Mary's Hospital, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Southwest Illinois Health Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - Mission Cancer and Blood - Ankeny, Ankeny, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Mission Cancer and Blood - West Des Moines, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mission Cancer and Blood - Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Mission Cancer and Blood - Laurel, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Saint Joseph Mount Sterling, Mount Sterling, Kentucky
  - Mercy Health - Paducah Medical Oncology and Hematology, Paducah, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Saint Agnes Hospital, Baltimore, Maryland
  - Hickman Cancer Center, Adrian, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - MU Health Care Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Lake Regional Hospital, Osage Beach, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - BJC Outpatient Center at Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Morristown Medical Center, Morristown, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Garnet Health Medical Center, Middletown, New York
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Mercy Health Perrysburg Cancer Center, Perrysburg, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Baker City, Baker City, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - Community Medical Center, Scranton, Pennsylvania
  - Geisinger Medical Oncology-Selinsgrove, Selinsgrove, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Memorial Hospital, Chattanooga, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - Sovah Health Martinsville, Martinsville, Virginia
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - West Virginia University Healthcare, Morgantown, West Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Mayo Clinic Health System Eau Claire Hospital-Luther Campus, Eau Claire, Wisconsin
  - Marshfield Medical Center - Ladysmith, Ladysmith, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Froedtert and MCW Moorland Reserve Health Center, New Berlin, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming